CLINICAL TRIAL: NCT04190810
Title: Mechanisms Underlying the Approach and Avoidance Task (AAT) in Smoking Cessation
Brief Title: The Approach and Avoidance Task (AAT) in Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAT002
Record Dates: First submitted 2019-08-11; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Smoking Cessation
Keywords: Approach and Avoidance Task (AAT); Inhibition; fMRI
MeSH Terms: conditions — Smoking Cessation; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Smokers, who just quitted smoking or start with smoking cessation, are randomly assigned to one of three conditions and are tested on three consecutive points in time.
Who Masked: Participant
Masking Description: Participants do not know that there exists more than one condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inhibition group (Experimental): The inhibition group gets the instructions to respond to pictures that are not related to smoking by swiping/pulling them towards themselves, whereas pictures with tobacco-related content shall be ignored. Up on pulling the pictures successively enlarge, whereas they shrink when ignored and slowly fade out.
  Interventions: Behavioral: Inhibition
- Classical AAT group (Experimental): The classical AAT group is provided with a tablet on which an explicit AAT training is installed. Thus, just as participants in the inhibition group, participants are instructed to react upon non-smoking related images by swiping/pulling towards themselves the picture. Pictures containing tobacco-related content shall be pushed away. Up on pulling pictures enlarge and up on pushing they shrink until they fade out.
  Interventions: Behavioral: Classical AAT
- Control group (Sham Comparator): This type of active control group receives the instructions to swipe tobacco-related pictures to the left and non-tobacco related pictures to the right (or vice versa depending on the sequential counterbalancing procedure).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Inhibition — Participants receive an Ipad, on which the app is installed. They are instructed to train for a period of three weeks for at least 15 minutes a day.
  Arms: Inhibition group
Behavioral: Classical AAT — Participants receive an Ipad, on which the app is installed. They are instructed to train for a period of three weeks for at least 15 minutes a day.
  Arms: Classical AAT group
Behavioral: Control — Participants receive an Ipad, on which the app is installed. They are instructed to train for a period of three weeks for at least 15 minutes a day.
  Arms: Control group

SUMMARY:
The approach and avoidance task (AAT) has evolved as a promising treatment add-on in the realm of psychology. Certain psychiatric diseases, such as behavioural addictions, social anxiety disorder, and arachnophobia, are characterized by a dysfunctional tendency to either approach or avoid disease-specific objects. This tendency can be measured by means of the approach and avoidance task. More precisely, by a diagnostic AAT, in which participants are instructed to react upon the format or the frame colour of a picture. For instance, pictures have to be pushed away if they are presented in landscape format and pulled towards oneself if they are presented in portrait format (or vice versa). Hence, the format (or the frame colour) becomes the task-relevant dimension, whereas the content of the picture becomes irrelevant for task completion. However, what generally becomes obvious in the psychiatric diseases mentioned above is that the task-irrelevant dimension (picture content) exerts an influence on reaction times. For instance, smokers are generally faster to respond to smoking-related pictures, when presented in a format requiring them to pull towards themselves, and slower to respond, if smoking pictures are shown in the format requiring them to push away a joystick (Wiers et al., 2013). This behavioural tendency has been termed an approach bias for cigarettes or smoking.

In order to counteract these dysfunctional approach or avoidance tendencies, an AAT-training has been developed. In this training participants/patients learn to either avoid or approach disease-specific objects. Smokers, for instance, learn to avoid smoking-related pictures by pushing or swiping the image away. It has been shown that these trainings can lower cigarette consumption among current smokers (Machulska, Zlomuzica, Rinck, Assian, & Margraf, 2016). The aim of the current study is to test whether the avoidance gesture is as important as suggested by the AAT's name or whether inhibiting the urge to approach smoking-related content might be enough to bring about the effect. Furthermore, possible changes in general and domain-specific (i.e. smoking-related) inhibition capacity, that might mediate the effect, will be assessed. Another focus of study will be on functional as well as structural neuronal changes, emerging as a consequence of the AAT-training.

DETAILED DESCRIPTION:
The approach and avoidance task (AAT) has turned out as both a promising diagnostic tool as well as treatment add-on in psychological science. The AAT constitutes one form of cognitive bias modification (CBM), which has been shown to be particularly effective in the field of behavioural addictions (Eberl et al., 2013; Wiers, Eberl, Rinck, Becker, & Lindenmeyer, 2011). The general logic underlying the AAT is to carry out actions that are either compatible or incompatible with an individual's action tendencies. For instance, nicotine addicted individuals tend to approach tobacco-related stimuli faster than control pictures, when they are instructed to react upon the format of a picture and not to its' content. This tendency of comparatively faster approaching and slower avoiding tobacco-related content has been termed an approach bias nicotine/tobacco. The AAT as a therapeutic tool tries to counteract or at least to attenuate approach or avoidance biases by instructing patients to carry out approach or avoidance gestures that are in conflict with an individual's acquired action tendencies.

Whereas the general effectiveness of the AAT as a clinical intervention has been demonstrated several times, little is known about possible mechanisms that might subserve these effects. Therefore, the current study is dedicated to shed some light on one such potential mechanism, i.e. the role of the avoidance gesture within the alcohol-AAT.

As already suggested by the name of the AAT, the avoidance gesture seems to be a key ingredient in bringing about therapeutic effects. However, recent empirical evidence has brought about some interesting findings, giving rise to an alternative explanation.

A study by Kühn et al. (2017), contrary to common-held beliefs, indicated that inhibition capacity can be trained. Inhibition, in turn, consistently has been linked to psychopathology and all kinds of behavioural addictions (Smith, Mattick, Jamadar, & Iredale, 2014). The game by Kühn et al. (2017), used to train inhibition, resembled the AAT in several ways, e.g. certain stimuli appearing on a treadmill had to be collected by swiping towards oneself and others had to be ignored and the objects slowly disappeared. The latter element contrasts with the AAT, since the ignored objects don't have to be pushed away. However, it resembles the AAT in the sense that in both cases stimuli slowly fade out of the screen and eventually disappear. These parallel let to the assumption that a new form of the alcohol AAT training might be equally effective in lowering relapse rates among alcoholic patients. More precisely, within the newly conceptualized AAT training, patients are instructed to inhibit the urge to respond in response to alcohol-related content and to observe the stimuli fading out of the screen. In contrast to the classical AAT training, this zooming out of alcoholic stimuli is not conditional on the avoidance gesture, i.e. swiping/pushing away the stimulus.

It is hypothesized that compared to a control group, in which tobacco and control stimuli have to be swiped to the left and right, both the classical AAT-and the inhibition group will be more successful in stopping or reducing smoking. The intervention includes a training period of four weeks. No intergroup differences in terms of smoking cessation and tobacco-related approach bias are expected for the classical AAT group and the inhibition group after the intervention.

Furthermore, it will be explored whether inhibition capacity changes as a result of the intervention, the assumption being that inhibition capacity increases for both experimental groups, whereas no changes are expected for the control group. An interesting question concerns the domain-specificity of potential effects. In other words, does inhibition capacity improve only for the to be trained domain (i.e. tobacco) or does the general inhibition capacity improve, irrespective of the to be trained domain? Predictions on this issue are not straightforward, but it is assumed that both the general and domain-specific inhibition capacity improve for the experimental groups, when compared to the control group. Slightly more pronounced effects are expected for the domain-specific task, since the training calls for comparable skills.

Hypotheses concerning experimental changes in brain structure are hard to make, as, to the best of our knowledge, no research has been done on this topic up until now. Therefore, whole-brain analyses will be run on all voxels of the brain in order to explore any experimental changes both on the within and between subject level.

The same goes for functional changes in a Stop Signal Task (SST) and a cue reactivity paradigm. It will be explored whether the classical AAT group and the inhibition group show less reward-related activity in response to addiction-related stimuli than participants in the control group. Furthermore, it will be explored whether brain regions commonly associated with inhibition capacity show more activity in response to smoking-related stimuli, since this has been learned throughout the training period.

All secondary outcome measures (e.g. smoking-related questionnaires, Beck's Depression Inventory, Barratt's Impulsivity Scale, AUDIT) assess whether the experimental manipulations lead to a reduction in psychopathological symptoms. Therefore, both experimental groups are expected to show post-interventional declines in nicotine-dependence measures and other measures associated with dependence, such as mental well-being and impulsivity. In contrast, no changes across time are expected for the control group.

In order to test prior mentioned hypotheses, a randomized controlled trial will be conducted. Each of the three groups (inhibition group, classical AAT group, and control group) will consist out of 25 mentally healthy participants, who just stopped smoking or just start an attempt to quit smoking.

In total the study consists out of three points of measurement. After the baseline testing, which assesses participants' approach bias for tobacco, their tobacco history, tobacco consumption within the last months, a multitude of smoking-related questionnaires (see secondary outcome measures), the two inhibition tasks, brain structure and brain function, participants are provided with a tablet on which the AAT app is installed. The participants are asked to train with the app for at least 15 minutes daily within a four-week period. Following this training, the second point of measurement will take place. The general procedure is identical to the first point of measurement. Another four weeks later, the third point of measurement marks the end of the study. Once again, the measures are the same except for the fact that no MRI scan is realized on this last occasion, since the study is primarily interested in post-interventional brain changes.

ELIGIBILITY:
Inclusion Criteria:

* being mentally healthy
* just having stopped smoking or having the urge to do so
* adequate language skills
* being right-handed

Exclusion Criteria:

* MRI contra indications, such as claustrophobia, tinnitus, and having any non-removable ferromagnetic artefacts within the body
* somatic or neurological disease that precludes the proper execution of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Fagerström Test of Nicotine Dependence (FTND) | 2 months
  Fagerstrom test for nicotine addiction determines the degree of nicotine dependence based on smoking habits and frequency.
Number of cigarettes consumed within the last month | 2 months
  On each point of measurement the number of cigarettes that has been smoked during the last month will be assessed by means of a memory protocol.
Diagnostic AAT | 2 months
  Two diagnostic AAT scores will be assessed on each point of measurement. One on a tablet and the other employing a joystick and a computer. The sequence is the same across testing sessions for the respective participant, but will be randomly counterbalanced between participants.
Cigarette Dependence Scale | 2 months
  Measures the extent of nicotine dependence.
GoNoGo Task | 2 months
  Numbers 1-9 appear on the screen in random sequence. Participants are asked to respond as fast as possible by pushing the space bar on all trials except those showing the number 3. On these trials participants are asked to suppress, i.e. inhibit a response.
Stop Signal Task (SST) | 2 months
  Participants have to respond to pictures with blue and yellow frames by pressing a left and right computer key, respectively (or vice versa depending on counterbalancing). These key presses shall be executed as quick as possible, when pictures are presented. However, on certain trials an acoustic stop signal follows the presentation of the picture. On these trials participants are asked to inhibit their response, and hence not to press any key.

SECONDARY OUTCOMES:
Smoking Behavior of Meaningful Others (Questionnaire) | 2 months
  This questionnaire assesses both the smoking habits of meaningful others as well as their appraisal of the participants' smoking behavior
Cue Exposure Questionnaire | 2 months
  Measures the extent to which certain cues (situations or places) induce the urge to smoke a cigarette.
Questionnaire of Smoking Urges | 2 months
  Measures the current urge to smoke a cigarette.
Commitment to Quitting Smoking Scale | 2 months
  Assesses the motivation to stop/reduce smoking.
Obsessive Compulsive Smoking Scale | 2 months
  Measures the extent to which thoughts and actions are occupied by smoking urges.
Barratt Impulsiveness Scale | 2 months
  A questionnaire designed to assess the personality/behavioral construct of impulsiveness.
Beck's Depression Inventory | 2 months
  Assesses the degree of depressive symptoms.
Alcohol Use Disorders Identification Test (AUDIT) | 2 months
  The AUDIT is a simple method of screening for excessive drinking and alcohol use disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Kühn, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Clinic Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wiers CE, Kuhn S, Javadi AH, Korucuoglu O, Wiers RW, Walter H, Gallinat J, Bermpohl F. Automatic approach bias towards smoking cues is present in smokers but not in ex-smokers. Psychopharmacology (Berl). 2013 Sep;229(1):187-97. doi: 10.1007/s00213-013-3098-5. Epub 2013 Apr 19. PMID 23604335
- [Result] Machulska A, Zlomuzica A, Rinck M, Assion HJ, Margraf J. Approach bias modification in inpatient psychiatric smokers. J Psychiatr Res. 2016 May;76:44-51. doi: 10.1016/j.jpsychires.2015.11.015. Epub 2015 Dec 13. PMID 26874269
- [Result] Eberl C, Wiers RW, Pawelczack S, Rinck M, Becker ES, Lindenmeyer J. Approach bias modification in alcohol dependence: do clinical effects replicate and for whom does it work best? Dev Cogn Neurosci. 2013 Apr;4:38-51. doi: 10.1016/j.dcn.2012.11.002. Epub 2012 Nov 14. PMID 23218805
- [Result] Wiers RW, Eberl C, Rinck M, Becker ES, Lindenmeyer J. Retraining automatic action tendencies changes alcoholic patients' approach bias for alcohol and improves treatment outcome. Psychol Sci. 2011 Apr;22(4):490-7. doi: 10.1177/0956797611400615. Epub 2011 Mar 9. PMID 21389338
- [Result] Kuhn S, Lorenz RC, Weichenberger M, Becker M, Haesner M, O'Sullivan J, Steinert A, Steinhagen-Thiessen E, Brandhorst S, Bremer T, Gallinat J. Taking control! Structural and behavioural plasticity in response to game-based inhibition training in older adults. Neuroimage. 2017 Aug 1;156:199-206. doi: 10.1016/j.neuroimage.2017.05.026. Epub 2017 May 17. PMID 28527788
- [Result] Smith JL, Mattick RP, Jamadar SD, Iredale JM. Deficits in behavioural inhibition in substance abuse and addiction: a meta-analysis. Drug Alcohol Depend. 2014 Dec 1;145:1-33. doi: 10.1016/j.drugalcdep.2014.08.009. Epub 2014 Aug 24. PMID 25195081